CLINICAL TRIAL: NCT06862713
Title: Determination of the Effects of Walking and Home-Based Pulmonary Rehabilitation on Anxiety and Sleep Quality in Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial
Brief Title: Effects of Walking and Home-Based Pulmonary Rehabilitation on Anxiety and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bilecik12
Record Dates: First submitted 2025-02-11; First posted 2025-03-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; pulmonary rehabilitation; exercise; anxiety; sleep quality; randomized controlled trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Study Population and Sample The study population will consist of patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD) who visit the chest diseases outpatient clinic of a training and research hospital and meet the study criteria. In this study, the anxiety level in COPD patients is determined as the primary observational variable. A power analysis is planned to determine the sample size of the study. Before conducting the power analysis, the effect size will be estimated based on a similar study previously conducted in the literature. Based on this study, Type-1 error (α) = 0.05, power (1-β) = 0.90, and effect size calculated for the Student's t-test (d = 0.364) were determined. Based on these parameters, the minimum required sample size is expected to be 41 patients per group, with a total of 82 participants. However, considering potential losses during the study process, it is planned to include a total of 90 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): pulmonary rehabilitation exercise + standard protocol
  Interventions: Behavioral: pulmonary rehabilitation exercise
- Control group (No Intervention): standard protocol

INTERVENTIONS:
Behavioral: pulmonary rehabilitation exercise — pulmonary rehabilitation exercise + standard protocol
  Arms: Intervention group

SUMMARY:
Although pulmonary rehabilitation plays an important role in increasing exercise tolerance and reducing hospitalizations in patients with chronic obstructive pulmonary disease (COPD), adherence to treatment is often low. Therefore, home-based pulmonary rehabilitation (PR) programs stand out as an effective intervention to alleviate the physiological and psychological burden of COPD patients and improve their quality of life. Nursing should develop a holistic approach to addressing the physical and psychological needs of patients to enhance the effectiveness of these programs.

This study aims to evaluate the effects of an 8-week home-based PR program on cardiopulmonary parameters, respiratory function, anxiety levels, and sleep quality in COPD patients.

As a randomized controlled trial, COPD patients will be divided into experimental and control groups. Pre- and post-tests will include the 6-minute walking test (6 MWT), dyspnea score, oxygen saturation, respiratory function tests (FEV1, FVC, FEV1/FVC, FEF 25-75), anxiety (STAI-I and STAI-II), and sleep quality (PSQI). Post-tests will be collected after the eight-week intervention.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common, preventable, and treatable disease characterized by exposure to harmful agents, associated with increased chronic inflammatory response of the lung, causing shortness of breath and significant systemic effects. COPD symptoms include not only shortness of breath, chronic cough, and increased sputum production, but also decreased exercise tolerance.

Although there are various treatment options that can reduce COPD symptoms (smoking cessation, pharmacological treatment, vaccines, etc.), there is no treatment yet that can return lung functions to their pre-disease normal state. Therefore, pulmonary rehabilitation is an important scientifically based, safe, and effective non-pharmacological treatment option recommended in guidelines for COPD patients to maintain the patient's quality of life. The most important component of pulmonary rehabilitation in COPD is exercise training. Pulmonary rehabilitation has been shown to increase exercise tolerance in patients with COPD, reduce re-admissions to hospital, and improve health status. Home-based pulmonary rehabilitation stands out as an alternative model that can overcome these barriers and increase access and participation. Initial studies suggest that home-based PR is safe and may improve clinical outcomes. The effectiveness of pulmonary rehabilitation in COPD patients is directly related to the patient's compliance with the program.

Difficulties experienced due to COPD also negatively affect the psychosocial status of patients. Shortness of breath can trigger anxiety and panic attacks in COPD patients. Anxiety and depression can worsen the health status of COPD patients and cause increased morbidity. In a study was determined that exercise improves anxiety and depression symptoms in COPD patients and increases the quality of life of patients. In addition, patients often complain of chronic insomnia; nearly 50% of patients report difficulty falling asleep, staying asleep, or experiencing unrefreshing sleep. The fact that there is no study in our country on non-pharmacological methods (pulmonary rehabilitation and exercise) to improve both anxiety and sleep quality in COPD patients and that an individual-focused pulmonary rehabilitation training program has been designed reveals the importance of this study and its contribution to the literature. This study evaluates the effects of walking and home-based pulmonary rehabilitation programs on anxiety and sleep quality in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to speak and understand Turkish
* Baseline saturation > 85%
* Confirmed stage II or stage III COPD diagnosis according to GOLD guidelines
* No infection or COPD exacerbation in the last 3 months
* Not participating in a pulmonary rehabilitation program in the last 3 months
* Able to walk without assistance and lift weights up to 2 kg
* No history of serious and/or unstable heart disease, neuromuscular disease, orthopedic disease, or mental illness that may affect daily physical activities
* Agree to participate in the study and give written informed consent
* No communication problems

Exclusion Criteria:

* Patients who require hospitalization after starting the study
* Patients receiving continuous oxygen therapy
* Patients with a history of pulmonary hypertension, malignancy, pulmonary thromboembolism, obstructive sleep apnea, unstable angina, or myocardial infarction
* Patients with a heart rate above 120/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory (STAI-I and STAI-II) | At baseline (first visit) and at 8 weeks
  The Spielberger State-Trait Anxiety Inventory (STAI-I and STAI-II), developed by Spielberger et al. (1970) and adapted to Turkish by Öner and Le Compte (1995), assesses anxiety levels in individuals aged 14 and above. The inventory consists of two subscales, each with 20 items rated on a 4-point Likert scale.
  STAI-I (State Anxiety): Measures how an individual feels at a specific moment under certain conditions (1 = Not at all, 4 = Completely). STAI-II (Trait Anxiety): Evaluates the individual's general anxiety tendency in the absence of external threats (1 = Almost never, 4 = Almost always). Each subscale includes reverse-scored items (10 in STAI-I, 7 in STAI-II). Total scores range from 20 to 80, with higher scores indicating greater anxiety. The average scores typically range between 36 and 41.
Pittsburgh Sleep Quality Index (PSQI) | At baseline (first visit) and at 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI), assesses sleep quality and habits over the past month. The scale consists of 19 self-reported items and 5 additional items answered by a bed partner or roommate (not included in scoring).
  The PSQI includes seven components:
  Subjective sleep quality Sleep latency Sleep duration Habitual sleep efficiency Sleep disturbances Use of sleep medication Daytime dysfunction Each component is scored between 0 (best) and 3 (worst), with a total score ranging from 0 to 21. Higher scores indicate poorer sleep quality, and a total score above 5 is considered indicative of poor sleep quality. The PSQI does not diagnose sleep disorders but serves as a useful tool for evaluating overall sleep quality. The reliability analysis reported a Cronbach's α of 0.80.
6 Minute Walk Test (6MWT) Distance | At baseline (first visit) and at 8 weeks
  Distance walked (meters) in the 6-Minute Walk Test. Higher distance indicates better functional capacity.
Modified Borg Dyspnea Scale (MBS) | At baseline (first visit) and at 8 weeks
  The Modified Borg Scale (MBS) assess perceived exertion during physical activity. It is one of the most reliable scales for evaluating dyspnea severity during both rest and exertion.The MBS consists of 10 items, each describing increasing levels of dyspnea intensity. It is simple to use and has been shown to correlate with pulmonary function tests. Dyspnea is assessed using the MBS at the end of the 6-Minute Walk Test (6MWT).
  The scale ranges from 0 (no breathlessness) to 10 (maximum breathlessness).
Pulmonary Function Tests (FEV1) | At baseline (first visit) and at 8 weeks
  Forced expiratory volume in 1 second (FEV1), Unit of Measure: percent (%), Higher FEV1 percentile is associated with better respiratory function.
Oxygen Saturation (SpO2, %) at Rest | At baseline (first visit) and at 8 weeks
  Oxygen saturation (%) will be measured using a pulse oximeter at rest. Higher values indicate better oxygenation.
Pulmonary Function Tests (FVC) | At baseline (first visit) and at 8 weeks
  Forced vital capacity (FVC), Unit of Measure: percent (%), Higher FVC percentile is associated with better respiratory function.
Pulmonary Function Tests (FEV1/FVC) | At baseline (first visit) and at 8 weeks
  The FEV1/FVC ratio is the ratio of the patient's forced expiratory volume in the first 1 second to the total mandatory vital capacity. FEV1/FVC ratio will be measured using spirometry. Unit of Measure: percent (%), Higher FEV1/FVC percentile is associated with better respiratory function.
Pulmonary Function Tests (FEF25-75%) | At baseline (first visit) and at 8 weeks
  Forced expiratory flow rate (FEF25-75%) represents the midairway flow rate between 25% and 75% of forced expiration. Unit of Measure: percent (%).An increase in FEF 25-75% may indicate improvement in small airways and a decrease in obstructive airway diseases.

CONTACTS AND LOCATIONS:
Overall Officials: SABAHAT COŞKUN, Doç.Dr., Study Director — Bilecik Şeyh Edebali Üniversity
Locations (1):
- Gulhane Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request, in accordance with ethical guidelines and with participant consent.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Xu J, He S, Han Y, Pan J, Cao L. Effects of modified pulmonary rehabilitation on patients with moderate to severe chronic obstructive pulmonary disease: A randomized controlled trail. Int J Nurs Sci. 2017 Jun 27;4(3):219-224. doi: 10.1016/j.ijnss.2017.06.011. eCollection 2017 Jul 10. PMID 31406744
- [Background] Zhang Y, Li G, Liu C, Guan J, Zhang Y, Shi Z. Comparing the efficacy of different types of exercise for the treatment and prevention of depression in youths: a systematic review and network meta-analysis. Front Psychiatry. 2023 Jun 2;14:1199510. doi: 10.3389/fpsyt.2023.1199510. eCollection 2023. PMID 37333923
- [Background] Yang PY, Ho KH, Chen HC, Chien MY. Exercise training improves sleep quality in middle-aged and older adults with sleep problems: a systematic review. J Physiother. 2012;58(3):157-63. doi: 10.1016/S1836-9553(12)70106-6. PMID 22884182
- [Background] Soler X, Diaz-Piedra C, Ries AL. Pulmonary rehabilitation improves sleep quality in chronic lung disease. COPD. 2013 Apr;10(2):156-63. doi: 10.3109/15412555.2012.729622. Epub 2013 Mar 20. PMID 23514215
- [Background] Li M, An X, Wang Q, Ma J, Wang Y, Ma J. Effect of Hope Theory combined with active cycle of breathing techniques on pulmonary rehabilitation among COPD patients: A quasi-experiment study. Appl Nurs Res. 2024 Oct;79:151842. doi: 10.1016/j.apnr.2024.151842. Epub 2024 Aug 26. PMID 39256012
- [Background] Li J, Lu Y, Li N, Li P, Su J, Wang Z, Wang T, Yang Z, Yang Y, Chen H, Xiao L, Duan H, Wu W, Liu X. Muscle metabolomics analysis reveals potential biomarkers of exercise-dependent improvement of the diaphragm function in chronic obstructive pulmonary disease. Int J Mol Med. 2020 Jun;45(6):1644-1660. doi: 10.3892/ijmm.2020.4537. Epub 2020 Mar 12. PMID 32186768
- [Background] Cox NS, Pepin V, Burge AT, Hill CJ, Lee AL, Bondarenko J, Moore R, Nicolson C, Lahham A, Parwanta Z, McDonald CF, Holland AE. Pulmonary Rehabilitation does not Improve Objective Measures of Sleep Quality in People with Chronic Obstructive Pulmonary Disease. COPD. 2019 Feb;16(1):25-29. doi: 10.1080/15412555.2019.1567701. Epub 2019 Mar 19. PMID 30884984
- [Background] Higginson R, Parry A. Managing chronic obstructive pulmonary disease in the community setting. Br J Community Nurs. 2018 Jan 2;23(1):6-12. doi: 10.12968/bjcn.2018.23.1.6. PMID 29281912
- [Background] Bains D, Chahal A, Shaphe MA, Kashoo FZ, Ali T, Alghadir AH, Khan M. Effects of Muscle Energy Technique and Joint Manipulation on Pulmonary Functions, Mobility, Disease Exacerbations, and Health-Related Quality of Life in Chronic Obstructive Pulmonary Disease Patients: A Quasiexperimental Study. Biomed Res Int. 2022 Jul 30;2022:5528724. doi: 10.1155/2022/5528724. eCollection 2022. PMID 35941972
- [Background] Alnawwar MA, Alraddadi MI, Algethmi RA, Salem GA, Salem MA, Alharbi AA. The Effect of Physical Activity on Sleep Quality and Sleep Disorder: A Systematic Review. Cureus. 2023 Aug 16;15(8):e43595. doi: 10.7759/cureus.43595. eCollection 2023 Aug. PMID 37719583
- [Background] Aiello M, Frizzelli A, Pisi R, Accogli R, Marchese A, Carlacci F, Bondarenko O, Tzani P, Chetta A. Effects of Daily Physical Activity on Exercise Capacity in Chronic Obstructive Pulmonary Disease. Medicina (Kaunas). 2024 Jun 21;60(7):1026. doi: 10.3390/medicina60071026. PMID 39064455
- [Background] Adeloye D, Agarwal D, Barnes PJ, Bonay M, van Boven JF, Bryant J, Caramori G, Dockrell D, D'Urzo A, Ekstrom M, Erhabor G, Esteban C, Greene CM, Hurst J, Juvekar S, Khoo EM, Ko FW, Lipworth B, Lopez-Campos JL, Maddocks M, Mannino DM, Martinez FJ, Martinez-Garcia MA, McNamara RJ, Miravitlles M, Pinnock H, Pooler A, Quint JK, Schwarz P, Slavich GM, Song P, Tai A, Watz H, Wedzicha JA, Williams MC, Campbell H, Sheikh A, Rudan I. Research priorities to address the global burden of chronic obstructive pulmonary disease (COPD) in the next decade. J Glob Health. 2021 Oct 9;11:15003. doi: 10.7189/jogh.11.15003. eCollection 2021. PMID 34737870
- [Derived] Coskun S, Simsek NY, Arslan Y. Effects of Home-Based Pulmonary Rehabilitation on Walking, Anxiety and Sleep in Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Int J Nurs Pract. 2025 Dec;31(6):e70085. doi: 10.1111/ijn.70085. PMID 41351250